CLINICAL TRIAL: NCT01444716
Title: Phase II Study of Ofatumumab as Front-Line Treatment in Elderly, Unfit Patients With Chronic Lymphocytic Leukemia (CLL)
Brief Title: Ofatumumab as Front-Line Therapy in Treating Elderly Participants With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0520; NCI-2018-01841 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2011-0520 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2011-09-28; First posted 2011-10-03 (Estimated); Results first posted 2021-07-26 (Actual); Last update posted 2021-07-26 (Actual); Status verified 2021-07

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ofatumumab) (Experimental): Participants receive ofatumumab IV over 4 hours once a week for 4 weeks, then monthly thereafter. Treatment continues for up to 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ofatumumab

INTERVENTIONS:
Biological: Ofatumumab — Given IV
  Other Names: Arzerra; GSK1841157; HuMax-CD20; HuMax-CD20, 2F2

SUMMARY:
This phase II trial studies how well ofatumumab works as front-line therapy in treating elderly participants with chronic lymphocytic leukemia. Monoclonal antibodies, such as ofatumumab, may interfere with the ability of cancer cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES I. To evaluate the overall response rate of ofatumumab in the upfront setting in elderly, unfit patients with chronic lymphocytic leukemia (CLL).

SECONDARY OBJECTIVES:

I. To determine the overall survival with ofatumumab in upfront setting in elderly, unfit CLL patients.

II. To evaluate the complete response rate and time to progression to therapy of ofatumumab in elderly, unfit patients with CLL.

III. To determine the plasma levels of ofatumumab in elderly, unfit patients. IV. To evaluate predictive capability of micro ribonucleic acid (RNA) (miRNAs) detection in plasma samples.

OUTLINE:

Participants receive ofatumumab intravenously (IV) over 4 hours once a week for 4 weeks, then monthly thereafter. Treatment continues for up to 12 months in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic lymphocytic leukemia requiring treatment at the time of signing informed consent.
* Eastern Cooperative Oncology Group (ECOG)/World Health Organization (WHO) performance status of 2-3 and a Cumulative Illness Rating Scale (CIRS) or Charlson co-morbidity score of 2 or higher.
* Creatinine < 2mg/dL.
* Estimated glomerular filtration rate (eGFR) more than 30cc/minute.
* Bilirubin < 2mg/dL.
* Patients with renal or liver dysfunction due to organ infiltration by lymphocytes may be eligible after discussion with the study chairman.
* Patients with Gilbert's syndrome are eligible.

Exclusion Criteria:

* Patients with documented prolymphocytic leukemia (prolymphocytes more than 55% in the blood).
* Known positivity for human immunodeficiency virus (HIV).
* Hepatitis B (HB) defined as a positive test for hepatitis B surface antigen (HBsAg). In addition, if negative for HGsAg but hepatitis B core antibody (HBcAb) positive (regardless of HBsAb status), a HB deoxyribonucleic acid (DNA) test will be performed and if positive the subject will be excluded.
* Prior treatment for chronic lymphocytic leukemia.
* Concurrent chemotherapy, radiotherapy, or immunotherapy, including other monoclonal antibodies. Localized radiotherapy to an area not compromising bone marrow function does not apply. Patients with malignancies with indolent behavior such as prostate cancer treated with radiation or surgery can be enrolled in the study as long as they have a reasonable expectation to have been cured with the treatment modality received.
* Any serious medical condition, laboratory abnormality, or psychiatric illness that places the subject at unacceptable risk if he/she were to participate in the study.
* Any known hypersensitivity to ofatumumab or its components.

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-12-15 (Actual); Primary Completion 2020-06-11 (Actual); Study Completion 2020-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Ferrajoli, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Ofatumumab)
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ofatumumab)
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 34
Age, Continuous [Median (Full Range); unit: years] | 73 [65 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 28
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Participants With a Response
Description: Response = (complete response [CR] + partial response [PR]) per 2008 National Cancer Institute (NCI)-Working Group (WG) criteria. Complete Response (CR): Absence of disease signs/symptoms, normalization of peripheral blood and bone marrow. Partial Response (PR): At least 50 % reduction in disease signs/symptoms and normalization of peripheral blood.
Time Frame: Up to 3 years, 10 months
Population: Of the 34 participants registered, 32 were evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ofatumumab)
Number analyzed (Participants) | 32
Participants | 23

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Time from date of treatment start until the date of first objective documentation of disease-relapse.
Time Frame: Up to 3 years, 10 months
Population: Of the 34 participants registered, 32 were evaluable for response.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Ofatumumab)
Number analyzed (Participants) | 32
Months | 21 [9 to 32]

3. Secondary Outcome: Participants With a Complete Response (CR)
Description: Complete Response (CR): Absence of disease signs/symptoms, normalization of peripheral blood and bone marrow.
Time Frame: Up to 3 years, 10 months
Population: Of the 34 participants registered, 32 were evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Ofatumumab)
Number analyzed (Participants) | 32
Participants | 6

ADVERSE EVENTS:
Time Frame: Up to 3 years, 10 Months
Arm/Group | Treatment (Ofatumumab)
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 9/34
Other Adverse Events (participants affected / at risk) | 29/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ofatumumab) (N=34)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Papillary Urothelial Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Transient Ichemic Attack (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Aortic Valve Disease (Cardiac disorders) | 1 (1)
Fever (General disorders) | 1 (2)
Lung Infection (Infections and infestations) | 1 (1)
Thromboembolic Event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ofatumumab) (N=34)
Abdoninal Pain (General disorders) | 7 (7)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Bone Fracture (Injury, poisoning and procedural complications) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Dizziness (Nervous system disorders) | 2 (2)
edema (General disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Fatigue (General disorders) | 5 (5)
Fever (General disorders) | 6 (6)
Headache (Nervous system disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 3 (3)
Infusion Related Reaction (General disorders) | 18 (19)
Mucositis (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Other Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Pain (General disorders) | 7 (7)
Palpitations (Cardiac disorders) | 2 (2)
Paresthesia (Nervous system disorders) | 3 (3)
Skin rash (Skin and subcutaneous tissue disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)
Infections (Infections and infestations) | 6 (7)
Skin Infection (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2)
Upper Respiratory Infection (Infections and infestations) | 7 (7)
Urinary Tract Infection (Infections and infestations) | 6 (6)
Urinary Incontinence (Renal and urinary disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-02-27): https://cdn.clinicaltrials.gov/large-docs/16/NCT01444716/Prot_SAP_000.pdf